CLINICAL TRIAL: NCT06306937
Title: Serum Levels of Vitamin D and IL8 in Patients With Periodontitis: A Case-control Study
Brief Title: Serum Levels of Vitamin D and IL8 in Patients With Periodontitis
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Wafaa Saleh, Assistant professor, Mansoura University
Other Study IDs: A24020822
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This study focuses on serum samples as the primary biospecimen, collected aseptically from individuals with and without periodontitis. Samples are meticulously labeled, processed through clotting and centrifugation, and stored at controlled temperatures in a secure bio-repository. The laboratory analysis will measure IL8 and vitamin D levels using standardized techniques. Each biospecimen is linked to participant data for correlation analysis, ensuring the integrity and confidentiality of the study's biospecimen collection and analysis process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis: Individuals diagnosed with periodontitis based on established clinical criteria. This group will include participants who exhibit signs and symptoms of periodontal disease, such as probing depth, clinical attachment loss, and bleeding on probing.
  Interventions: Diagnostic Test: Evalution of serum levels of vitamin D and IL8
- Control: Individuals without any signs or history of periodontal disease. This group will consist of participants who do not have clinically diagnosed periodontitis and serve as the healthy control group for comparison with the periodontitis group.
  Interventions: Diagnostic Test: Evalution of serum levels of vitamin D and IL8

INTERVENTIONS:
Diagnostic Test: Evalution of serum levels of vitamin D and IL8 — Group 1 (Periodontitis Group): The intervention involves observing and analyzing individuals diagnosed with periodontitis based on established clinical criteria. The focus is on assessing vitamin D and IL8 levels in the serum and correlating these levels with the severity of periodontitis, determined by clinical indices such as probing depth, clinical attachment loss, and bleeding on probing.
  Group 2 (Control Group): The intervention involves observing and analyzing individuals without any signs or history of periodontal disease. The focus is on assessing vitamin D and IL8 levels in the serum for comparison with the periodontitis group. This group serves as the healthy control for the study.

SUMMARY:
We evaluated vitamin D and IL8 levels in the serum of patients with periodontitis as well as the healthy controls to correlate their levels with the degree of periodontitis.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the levels of vitamin D and IL8 in the serum of individuals diagnosed with periodontitis and compare them with those of a healthy control group. The study also aims to establish correlations between these serum levels and the degree of periodontitis severity.

Two groups will be recruited: patients diagnosed with periodontitis and a control group consisting of individuals without periodontal disease.

The participants will be matched for age, gender, and other relevant demographic factors to minimize confounding variables.

Serum samples will be collected from both groups. Periodontitis severity will be determined using established clinical indices, such as probing depth, clinical attachment loss, and bleeding on probing.

Vitamin D levels in the serum will be measured using standardized laboratory techniques.

IL8 levels in the serum will also be quantified using appropriate assays. Statistical analyses will be performed to identify any significant correlations between vitamin D levels, IL8 levels, and the severity of periodontitis.

Subgroup analyses may be conducted to explore potential variations based on demographic factors or other relevant variables.

The study will adhere to ethical guidelines, ensuring participant confidentiality, informed consent, and responsible data handling.

The study anticipates finding associations or correlations between serum levels of vitamin D and IL8 and the severity of periodontitis. This information may contribute to a better understanding of the role of these factors in periodontal health and could have implications for future preventive and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least twenty teeth.
* Periodontitis patients with a minimum of 40% of sites with a clinical attachment level (CAL) ≥2 mm and probing depth (PD)≥4 mm.
* presence of ≥40% sites with bleeding on probing.
* Healthy individuals matched for age and gender, who presented no systemic disease, no drugs were taken, no sites with PD ≥4 mm or CAL ≥4 mm, or radiographic signs of bone loss were enrolled, such as a control group.

Exclusion criteria

* Intake of contraceptives, immunosuppressive, antibiotics or anti-inflammatory drugs throughout the last three months prior to the study.
* Pregnant and lactating females.
* Diabetic patients.
* History of medications that might affect bone and mineral metabolism and/or periodontal health.
* Taking multivitamins and food supplement which contain vitamin D.
* Malabsorption syndrome or patient with chronic diarrhea.
* Treatment with bisphosphonates in the past 12 months or lifetime exposure to bisphosphonates for more than 3 years.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Periodontitis Group: Individuals diagnosed with periodontitis, meet specific criteria such as a minimum of 40% of sites with CAL ≥2 mm, PD ≥4 mm, and ≥40% of sites with bleeding on probing. This group represented individuals with varying degrees of periodontal disease.
  Control Group: Healthy individuals, age, and gender-matched, devoid of systemic diseases, and medications, and with no sites exhibiting PD ≥4 mm or CAL ≥4 mm. This group provided a baseline for periodontal health in the absence of diagnosed periodontitis.
  The study's observational design allowed for the comprehensive examination of these groups, shedding light on the interplay between serum biomarkers, vitamin D, IL8, and periodontal health in a real-world setting. Population diversity enhances the generalizability of findings beyond specific clinical or demographic subsets.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Serum Levels of 25(OH)vitamin D | Laboratory evaluation after samples collection. it was performed in 1 month
  Measurement of vitamin D levels (categorized as deficient, inadequate, or adequate) using a commercial ELISA kit.
Serum Levels of IL8 | Laboratory evaluation after samples collection. it was performed in 1 month
  Measurement of IL8 levels (expressed in pg/ml) using a commercial ELISA kit.

SECONDARY OUTCOMES:
Plaque Index (Pl) | 1 day (Periodontal evaluation was performed one time for every patient with withdrawal of blood sample)
  Assessment of dental plaque presence and severity on a scale of 0 to 3.
Clinical Attachment Loss (CAL) | 1 day (Periodontal evaluation was performed one time for every patient with withdrawal of blood sample)
  Measurement in millimeters from CEJ to the most apically probable portion.
Probing Pocket Depth (PPD) | 1 day (Periodontal evaluation was performed one time for every patient with withdrawal of blood sample)
  Measurement in millimeters from the gingival margin to the most apically probable portion.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa saleh, Ph.D, Principal Investigator — Mansoura University, Faculty of Dentistry
Locations (1):
- Mansoura University, Faculty of Dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No